CLINICAL TRIAL: NCT03501940
Title: 18F-DCFPyL PET/CT in the Evaluation of Patients With Biochemical Recurrence of Prostate Cancer and Non-Contributory CT Scans
Brief Title: F18 DCFPyL PET/CT in Imaging Participants With Recurrent Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Andrei Iagaru (Other)
Responsible Party: Sponsor-Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Other Study IDs: IRB-42701; NCI-2018-00479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0083 (Other: OnCore)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Prostate Adenocarcinoma; PSA Level Greater Than 0.2; PSA Level Greater Than or Equal to Two; PSA Progression; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Procedure: Computed Tomography — Undergo 18F-DCFPyL PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fluorine F 18 DCFPyL — Given IV
  Other Names: 18F-DCFPyL
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo 18F-DCFPyL PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This study provides fluorine F 18 DCFPyL positron emission tomography/computed tomography (PET/CT) to participants with prostate cancer that has come back. Diagnostic procedures, such as fluorine F 18 DCFPyL PET/CT, may help find and diagnose prostate cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate fluorine F 18 DCFPyL (18F-DCFPyL) PET/CT for detection of recurrent prostate cancer after initial therapy in patients with elevated prostate-specific antigen (PSA).

OUTLINE:

Participants receive fluorine F 18 DCFPyL intravenously (IV). After 60-120 minutes, participants undergo whole body PET/CT. Immediately after the first scan, participants may undergo a second PET/CT without receiving fluorine F 18 DCFPyL.

After completion of study, participants are followed up at 24-72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma
* Rising PSA after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy)

  * Post radical prostatectomy (RP) - American Urological Association (AUA) recommendation

    * PSA greater than 0.2 ng/mL measured after at least 6 weeks from radical prostatectomy
    * Confirmatory persistent PSA greater than 0.2 ng/mL (total of two PSA measurements greater than 0.2 ng/mL)
  * Post-radiation therapy - American Society for Radiation Oncology (ASTRO) - Phoenix consensus definition

    * A rise of PSA measurement of 2 or more ng/mL over the nadir
* Able to provide written consent
* Karnofsky performance status of > 50 (or Eastern Cooperative Oncology Group [ECOG] / World Health Organization [WHO] equivalent)

Exclusion Criteria:

* Unable to provide informed consent
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

REFERENCES:
- [Derived] Baratto L, Song H, Duan H, Hatami N, Bagshaw HP, Buyyounouski M, Hancock S, Shah S, Srinivas S, Swift P, Moradi F, Davidzon G, Iagaru A. PSMA- and GRPR-Targeted PET: Results from 50 Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2021 Nov;62(11):1545-1549. doi: 10.2967/jnumed.120.259630. Epub 2021 Mar 5. PMID 33674398